CLINICAL TRIAL: NCT05141656
Title: Construction and Evaluation of China's Advanced Pancreatic Tumor Big Data Center
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CPOG-CDPC-01
Record Dates: First submitted 2021-11-20; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: Patients diagnosed as pancreatic tumor will considered to be enrolled regardless of specific pathologic subtypes expect for metastasis of pancreas. Baseline data and treatment information will be collected under fully informed consent.
  Interventions: Other: No intervention will be considered in this study.

INTERVENTIONS:
Other: No intervention will be considered in this study. — No intervention will be considered in this study.

SUMMARY:
This study is a multi-center observational study. The start time for data collection is August 31, 2019. Patients who have been treated at our institution from August 31, 2019, who were diagnosed with pancreatic tumors on or before August 31, 2019 (diagnosed in our hospital or outside hospitals) would all meet the inclusion conditions of the study and be considered enrollment. Patients' baseline and treatment data will be collected under informed concent. The combination of medical big data governance and the leading technology of the big data platform uses real world data to improve the quality and efficiency of pancreatic tumor diagnosis, treatment and scientific research.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, both male and female;
2. Patients with primary pancreatic tumor diagnosed by histology, cytology or imaging;
3. Clinical or pathological staging is locally advanced or metastatic pancreatic tumor (newly diagnosed or after surgery and other treatments);
4. You can accept or have not received surgery, chemotherapy, radiotherapy, local treatment or traditional Chinese medicine for tumors;
5. The subject voluntarily joined the study and signed an informed consent form voluntarily.

Exclusion Criteria:

1. Pancreatic tumors are evaluated as metastatic lesions, not primary tumors of the pancreas.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as tumor of pancreas will all be considered for enrollment.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-08-31 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
OS | 5 years
  overall survival

SECONDARY OUTCOMES:
DFS | 5 years
  disease free survival
PFS | 5 years
  progress free survival

CONTACTS AND LOCATIONS:
Locations (1):
- RenJiH, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided